CLINICAL TRIAL: NCT00307905
Title: A Randomised, Double - Blind, Placebo Controlled Clinical Trial to Assess the Efficacy of the Homeopathic Medication TRAUMEEL S in Controlling Post-operative Pain After Fracture of Neck of Femur
Brief Title: TRAUMEEL for Pain After Fracture of Neck of Femur
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Anticipation of inadequate recruitment according to current format.
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Menachem Oberbaum, MD, Shaare Zedek Medical Center,
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NoF 06 CTIL
Record Dates: First submitted 2006-03-27; First posted 2006-03-28 (Estimated); Last update posted 2010-10-29 (Estimated); Status verified 2010-10

CONDITIONS: Pain; Fracture of Neck of Femur
Keywords: homeopathy; pain; traumeel s; Fracture of neck of femur; Surgical correction of fracture of neck of hip
MeSH Terms: conditions — Pain; Femoral Neck Fractures | interventions — Traumeel S

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- A (Active Comparator): TRAUMEEL S
  Interventions: Drug: Traumeel S
- B (Placebo Comparator): placebo remedy
  Interventions: Drug: Placebo remedy

INTERVENTIONS:
Drug: Traumeel S — homeopathic remedy
  Arms: A
Drug: Placebo remedy — identical size, shape and taste of treatment medication
  Arms: B

SUMMARY:
We hypothesize that Traumeel S is more effective than placebo in reducing 48-hour mean cumulative morphine consumption in patients scheduled for surgical correction of fracture of neck of hip.

224 patients, meeting all inclusion and none of exclusion criteria, will be enrolled in the trial. Patients will be randomized to receive either intraoperative injection and post operative oral Traumeel S Tablets or placebo injection (normal saline) and indistinguishable oral placebo tablets. Baseline measurements of relevant outcome measures will taken preoperatively. Immediately after surgery, patients will receive an initial dose of morphine of 0.1mg/kg body weight. Patients will take the oral study medication for 21 days. Every four hours after surgery, patients will be asked to grade their pain on an NRS. Subsequent doses of morphine will be calculated based upon the patient's weight and current NRS, according to a preplanned scheme. Patients will be permitted to request additional morphine, beyond their calculated dose.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either sex undergoing surgical correction of unilateral fracture of neck of hip.
* Age over 18 years.
* Signature upon informed consent form

Exclusion Criteria:

* Participation in another clinical trial within 4 weeks prior to enrollment.
* Refused to give verbal consent to the telephone interviews
* Impossibility to be reached during the 14-17 days post operative
* Inability to comply with the study protocol for any other reason
* Previous major surgical procedure on ipsilateral hip.
* Current use of analgesics for any other reason.
* A history of chronic pain syndrome.
* Abused legal or illicit drug use.
* Hypersensitivity to botanicals of the Compositae family
* Known sensitivity to paracetamol, codeine or tramadol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Cumulative 48-hour postoperative morphine consumption | 48h

SECONDARY OUTCOMES:
Secondary: AUC of NRS scores for first 48 hrs.; | 48h
AUC of NRS scores for days 14-17.; | 17d
Composite measure of pain intensity and opiate consumption; | 17d
Number of primary oral analgesic tablets ingested between days 14-17; | 17d
ESR and hs-CPR at three and six days and six weeks; | 42d
IL-6 at three and six days; | 6d
Post operative blood loss; | 48h
WOMAC; | 17d
Safety of post operative treatment | 17d

CONTACTS AND LOCATIONS:
Overall Officials: Menachem Oberbaum, MD, Principal Investigator — Shaare Zedek Medical Center, Jerusalem, Israel
Locations (1):
- Dept. of Orthopedic Surgery, Shaare Zedek Medical Center, Jerusalem, Israel